CLINICAL TRIAL: NCT01687842
Title: Social Cognition and Turner Syndrome
Acronym: COGNITUR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110911; ID RCB 2012-A00488-35 (Other: ID RCB)
Record Dates: First submitted 2012-09-06; First posted 2012-09-19 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-10

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal DNA samples will be collected in the patient and her mother
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Turner syndrome patients: Evaluation of 45,X Turner syndrome patients
  Interventions: Other: Evaluation of 45,X Turner syndrome patients

INTERVENTIONS:
Other: Evaluation of 45,X Turner syndrome patients — Evaluation of 45,X Turner syndrome patients

SUMMARY:
Monocentric multidisciplinary study (psychologists, endocrinologists, psychiatrists, and molecular biologists) to characterize social cognition in adolescents with Turner syndrome (TS).

Inclusion criteria:

* Turner syndrome with homogeneous 45,X karyotype.
* Age between 8 and 18 years.
* Somatic state compatible with the evaluation.
* Functional language and IQ ≥ 80 for the transfer tests
* Informed consent signed by the holders of parental authority, the patient and the mother for her own participation (DNA collection).
* Affiliation to Social Security (beneficiary or assignee).

The primary endpoint will be the overall score to the AQ (Autism Quotient) questionnaire and to the SRS (Social Reciprocity Scale), in comparison to the expected scores for the general population. For patients with scores above the threshold for SRS or QA validation of a possible diagnosis of autism spectrum disorders will be performed with commonly used diagnostic tools (ADIR (Lord et al, 1994), ADOS-G (Lord et al, 1999) and diagnostic criteria of DSM IV-TR).

Secondary criteria will include the results of standardized tests to assess autistic features (AQ, ADI-R, ADOS, DSM IV-TR criteria), intellectual efficiency (Wechsler scales), psychiatric comorbidities (Kiddie-SADS) and sociocognitive profile (SpeX test, Social cognition, Perception, eXecutive functions).

A DNA sample will be collected from the patient and her mother. The observation period is 2 days for the patient and about 1 hour for the mother. The total duration of the study is 3 years.

DETAILED DESCRIPTION:
Patients will be recruited to the study by their pediatric endocrinologist during routine monitoring visits. They will then be contacted by phone or by mail for an appointment with their mother for more oral and written information consisting of an information notice and informed consent form. The recruitment of Turner syndrome patients will be based on the Reference Centre for Rare Endocrine Growth Disorders (AP-HP, Robert Debré, Armand Trousseau and Necker hospitals).

The parental origin of the remaining X chromosome will be analyzed using microsatellite analysis and comparison of the profile of the patient and her mother.

Statistical analysis will be conducted under the supervision of Professor C. ALBERTI using commonly accepted standards. All tests will be bilateral. Given the exploratory nature of the study, a significance threshold of 10% will be used. Statistical analyzes will be performed using SAS software V 9.2.

ELIGIBILITY:
Inclusion criteria:

* Turner syndrome with homogeneous 45,X karyotype.
* Age between 8 and 18 years.
* Somatic state compatible with the evaluation.
* Functional language and IQ ≥ 80 for the transfer tests
* Informed consent signed by the holders of parental authority, the patient and the mother for her own participation (DNA collection).
* Affiliation to Social Security (beneficiary or assignee).

Exclusion Criteria:

* Additional condition associated with an autism spectrum disorder
* Turner syndrome not related to an homogeneous 45,X karyotype

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Turner syndrome patients
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall score to the AQ (Autism Quotient) questionnaire. | 2 days
SRS (Social Reciprocity Scale), in comparison to the expected scores for the general population. | 2 days

SECONDARY OUTCOMES:
Socio-cognitive profile and parent of origin of the intact X chromosome | 2 days
  Results of standardized tests to assess autistic features (AQ, ADI-R, ADOS, DSM IV-TR criteria), intellectual efficiency (Wechsler scales), psychiatric comorbidities (Kiddie-SADS) and sociocognitive profile (SpeX test, Social cognition, Perception, eXecutive functions).
  Parent of origin of the intact X chromosome and its relationship to the autistic features.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Carel, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Delorme Richard, PHD, Study Chair — APHP
Locations (1):
- Robert Debre Hospital, Paris, France